CLINICAL TRIAL: NCT02574910
Title: A Phase 1 Multi-Center Study to Assess the Efficacy and Safety of Abiraterone Acetate as Adjunctive Therapy in Pre-Pubescent Children With Classic 21-Hydroxylase Deficiency
Brief Title: Androgen Reduction in Congenital Adrenal Hyperplasia, Phase 1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been affected significantly by the COVID pandemic, drug supply/drug amendment, low recruitment interest, and FDA approval of another drug with the same indication, so this study has not met its primary endpoint data requirements.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Michigan (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Perrin C White, MD, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 112014-087; 1U01HD083493-01 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-10-14 (Estimated); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Abiraterone acetate 1 mg/kg/d (Experimental): Abiraterone acetate will be administered orally at a daily dose of 1 mg/kg for 7 days in addition to the standard of care treatment of hydrocortisone and fludrocortisone.
  Interventions: Drug: Abiraterone acetate
- Abiraterone acetate 2 mg/kg/d (Experimental): If the 1 mg/kg/d dosing does not result in androstenedione level normalization, abiraterone acetate will be administered orally at a daily dose of 2 mg/kg for 7 days in addition to the standard of care treatment of hydrocortisone and fludrocortisone.
  Interventions: Drug: Abiraterone acetate
- Abiraterone acetate 4 mg/kg/d (Experimental): If the 2 mg/kg/d dosing does not result in androstenedione level normalization, abiraterone acetate will be administered orally at a daily dose of 4 mg/kg for 7 days in addition to the standard of care treatment of hydrocortisone and fludrocortisone.
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Abiraterone acetate — This is a dose escalation study. Up to 3 successive cohorts of 8 subjects each will receive 7 days of 1, 2 or 4 mg/kg/d of abiraterone acetate, until 7/8 subjects have met the desired endpoint.
  Other Names: Zytiga

SUMMARY:
Children with congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency tend to have elevated circulating levels of androgens, which can accelerate skeletal maturation and adversely impact adult height. Additionally, these children require supraphysiologic doses of hydrocortisone to suppress secretion of adrenal androgen precursors, and this treatment can retard linear growth. This study seeks to use oral abiraterone acetate (Zytiga)as an adjunct to approved CAH therapy (oral hydrocortisone and fludrocortisone) for pre-pubescent children with classic 21-hydroxylase deficiency in order to reduce daily requirement of hydrocortisone. In this Phase 1 study, the investigators will determine the minimum effective dose of abiraterone acetate that normalizes androstenedione levels during the 7-day Treatment Period.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is an inherited inability to synthesize cortisol in the adrenal gland. More than 90% of cases are cause by deficiency of steroid 21-hydroxylase (CYP21, also termed CYP21A2, P450c21), which is a cytochrome P450 enzyme located in the endoplasmic reticulum. It catalyzes conversion of 17-hydroxyprogesterone (17-OHP) to 11-deoxycortisol, a precursor for cortisol, and progesterone to deoxycorticosterone, a precursor for aldosterone. Aldosterone deficiency may lead to salt wasting with consequent failure to thrive, hypovolemia, shock and if untreated, death in the first few weeks of life. Because patients cannot synthesize cortisol efficiently, the adrenal cortex is stimulated by corticotropin (ACTH) and overproduces cortisol precursors. Some of these precursors are diverted to sex hormone biosynthesis, which may cause signs of androgen excess including ambiguous genitalia in newborn females, rapid postnatal growth in both sexes, and accelerated skeletal maturation and decreased adult height. Patients require supraphysiologic replacement doses of glucocorticoids to suppress the adrenocorticotropic hormone (ACTH)-driven adrenal androgen synthesis. Excessive glucocorticoids are associated with excessive weight gain and slowing of linear growth. It would be desirable in pre-pubertal children to decrease the exposure to excess glucocorticoids while avoiding the adverse effects of inappropriate exposure to androgens. Abiraterone acetate is a prodrug of abiraterone, an irreversible inhibitor of 17α hydroxylase/C17, 20-lyase (cytochrome P450c17 [CYP17]), a key enzyme required for testosterone synthesis. This agent indeed suppresses adrenal androgen secretion in adult women. In this Phase 1 study, the investigators will determine the minimum effective dose of abiraterone acetate that normalizes androstenedione levels during the 7-day Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-pubescent girls (age 2 years [12 kg minimum] to 8 years inclusive; skeletal age <10 years) or boys (age 2 years [12 kg] to 9 years inclusive; skeletal age <11 years).
2. Confirmed classic 21-hydroxylase deficiency evident by genotype groups A, A1 or B or clinical course (e.g., adrenal crisis with documented hyperkalemia and hyponatremia, at diagnosis or during a later evaluation; ambiguous genitalia in females). Documentation of one or both parents' genotypes may be required to confirm the subject's genotype.
3. Requirement for standard of care fludrocortisone (any dose) and ≥10 mg/m2/day of hydrocortisone for at least 1 month prior to the study consent.
4. Morning serum androstenedione concentrations >1.5 x Upper limit normal (ULN) after 7 days of dosing with doses of hydrocortisone required for physiologic replacement.
5. At least one parent (or other legally acceptable representative) must sign the informed consent form before the performance of any study procedures, but both parents must sign if both have parental rights. Children who are capable of providing assent (typically 10 years of age and older) must sign an assent form before the performance of any study procedures

Exclusion Criteria:

1. Evidence of central puberty: Tanner Stage >2 for breast development in girls or testicular volume >4 mL in boys, or random luteinizing hormone (LH) >0.3 milli-international units (mIU)/mL. Subjects with pubic and/or axillary hair as the only sign of puberty onset will be allowed.
2. Current or history of hepatitis from any etiology, including history of active viral hepatitis A, B, or C.
3. Patients with baseline hepatic impairment are excluded from this trial. To be eligible for this protocol, patients must meet all of the following criteria:

   AST, ALT and Total bilirubin < ULN Albumin > lower limits of normal (LLN) No evidence of ascites No evidence of encephalopathy
4. Abnormalities of liver function developing during the study
5. Abnormal renal function tests, defined as blood urea nitrogen (BUN) or creatinine >1.5 ULN for age.
6. Significant anemia (hemoglobin < 12 g/dl). If documented to be due to iron deficiency, subjects may be rescreened 3 months after this has been treated.
7. Clinically significant abnormality in the 12-lead electrocardiogram (ECG)
8. A history of a malabsorption syndrome.
9. Evidence of active malignancy.
10. Serious or uncontrolled co-existent disease, including active or uncontrolled infection. Subjects may be rescreened after resolution of any such condition.
11. Concurrent medical condition or disease other than 21-hydroxylase deficiency that may interfere with linear growth or that requires concomitant therapy that is likely to interfere with study procedures or results.
12. Asthma or other condition requiring treatment with systemic corticosteroids within the past 3 months. Asthma treatment with inhaled corticosteroids is permitted.
13. Treatment with potentially hepatotoxic medications (statins); strong inhibitors of CYP3A4 (ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, indinavir, nelfinavir, voriconazole), or CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital). CYP2C8 substrates (rosiglitazone, pioglitazone, rapaglinide) and CYP2D6 substrates (dextromethorphan, thioridazine) should be avoided
14. Treatment with medications to affect puberty or synthesis of sex steroids, including gonadotropin releasing hormone agonists, aromatase inhibitors, or androgen receptor blockers (e.g., flutamide, spironolactone). However, a gonadotropin releasing hormone agonist may be started during the study for treatment-emergent central puberty without disqualifying the subject
15. Treatment with growth hormone at enrollment or during the course of the study.
16. Known allergies, hypersensitivity, or intolerance to abiraterone acetate or its excipients (refer to United States Prescribing Information).
17. Has received an investigational drug within 4 weeks of the planned first dose of study drug or is currently enrolled in an investigational interventional study.
18. Any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
19. Presence or history of cataracts.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perrin C White, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - National Institutes of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Children's Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data Safety Monitoring Board plan
Supporting Information: Study Protocol

REFERENCES:
- [Background] Auchus RJ, Buschur EO, Chang AY, Hammer GD, Ramm C, Madrigal D, Wang G, Gonzalez M, Xu XS, Smit JW, Jiao J, Yu MK. Abiraterone acetate to lower androgens in women with classic 21-hydroxylase deficiency. J Clin Endocrinol Metab. 2014 Aug;99(8):2763-70. doi: 10.1210/jc.2014-1258. Epub 2014 Apr 29. PMID 24780050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Started | 2 | 2 | 0
Completed | 2 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 mg dose level not reached
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d | Total
Number analyzed (Participants) | 2 | 2 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 4
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 5 [5 to 5] | 7 [5 to 9] |  | 6 [5 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 2 | 2 | 0 | 4
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Normalization of Serum Androstenedione Level
Description: The original primary endpoint was the dose of abiraterone acetate that normalized androstenedione to age-appropriate levels in 7/8 subjects after 7 days of treatment. However, an insufficient number of participants was enrolled to evaluate the primary endpoint. Therefore, we have instead presented the number of participants at each dose level who did normalize androstenedione to age-appropriate levels.
Time Frame: 7 days
Population: No subjects enrolled at 4 mg/kg/d
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 2 | 2 | 0
Participants | 0 | 1 | 0

2. Secondary Outcome: 17-hydroxyprogestoerone Levels
Description: Final lab results at Screening and V6. This outcome is not pre-specified in the protocol and was inadvertently added at the time of registration.
Time Frame: 7 days
Population: Due to early termination of this study and incomplete enrollment, the collected data are incomplete and limited. These collected samples will never be analyzed in the future. Due to quality issues with the resulting of 17-hydroxyprogestoerone, there is one per-protocol patient to report this result on.
Measure: Number; unit: ng/dL
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 1 | 0 | 0
ng/dL | -2790 |  |

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Abiraterone
Description: Sparse pharmacokinetic (PK) will be derived from peak and trough abiraterone levels.
Time Frame: 7 days
Population: The values for this outcome measurement were not collected and we have no data relating to PK to report because the collected samples were not processed for this outcome measure and will never be processed in the future as well.
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Sparse pharmacokinetic (PK) will be derived from peak and trough abiraterone levels.
Time Frame: 7 days
Population: as for outcome 3
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Dihydrotestosterone Levels
Description: Final lab results at Screening and V6. This was erroneously listed as a secondary outcome in PRS. We have changed the outcome measure type to "Other pre-specified." .
Time Frame: 7 days
Population: Due to early termination of this study and incomplete enrollment, the collected data are incomplete and limited, it is not considered valid to perform this outcome measure assessment and therefore unable to analyze and report it.
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Adverse Events
Description: Safety monitoring in Phase 1 will include liver function tests (AST, Alanine Aminotransferease (ALT), bilirubin) and possible mineralocorticoid effects (blood pressure, plasma renin).
Time Frame: 7 days
Population: No participants enrolled at the 4 mg/kg/d level.
Measure: Number; unit: events
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
Number analyzed (Participants) | 2 | 2 | 0
events | 6 | 1 |

ADVERSE EVENTS:
Time Frame: 60 days
Description: No subjects were enrolled at the 4 mg/kg/d dose level.
Arm/Group | Abiraterone acetate 1 mg/kg/d | Abiraterone acetate 2 mg/kg/d | Abiraterone acetate 4 mg/kg/d
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abiraterone acetate 1 mg/kg/d (N=2) | Abiraterone acetate 2 mg/kg/d (N=2) | Abiraterone acetate 4 mg/kg/d (N=0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was adversely impacted by study drug availability, requiring reformulation; by the COVID19 pandemic; by competing industry sponsored Phase 2-3 trials of tildacerfont and crinecerfont, which targeted the same outcome in the same population; and by the eventual FDA approval of crinecerfont.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02574910/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02574910/ICF_001.pdf